CLINICAL TRIAL: NCT00567684
Title: Pilot Study Assessing the Technical Efficacy of Computed Tomography Urography (CTU) vs Intravenous Urography (IVU) With Particular Focus on Patients at Risk of Urothelial Tumors
Brief Title: Computed Tomography Urography (CTU) vs Intravenous Urography (IVU) on Patients at Risk of Urothelial Tumors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-0381; NCI-2014-01374 (Registry Identifier: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Bladder Cancer
Keywords: Transitional Cell Carcinoma; Urothelial Cancer; Bladder Cancer; Computed Tomography Urography; CTU; Intravenous Urography; IVU; TCC; transitional cell carcinomas
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CTU + IVU (Experimental): CTU = Computed Tomography Urography + IVU = Intravenous Urography
  Interventions: Device: Computed Tomography Urography (CTU); Other: Intravenous Urography (IVU)

INTERVENTIONS:
Device: Computed Tomography Urography (CTU) — CTU performed at least a day before or after the IVU procedure.
  Other Names: CTU
Other: Intravenous Urography (IVU) — A routine IVU procedure performed prior to or after CTU.
  Other Names: IVU

SUMMARY:
The goal of this clinical research study is to use computed tomography urography (CTU) scans and intravenous urography (IVU) scans to check the status of urothelial cancer, in order to try to learn the level of effectiveness of possibly using CTU by itself in future patients.

DETAILED DESCRIPTION:
Background for the Study:

Currently, IVU is used to detect urothelial tumors and then computed tomography (CT) scans are performed after that, to check the status of the disease. This is typically done every 3 months for the first 2 years after diagnosis, and then every 6 months for the next 2 years. Researchers want to learn if this current routine method of using 2 diagnostic procedures can be replaced with CTU alone, in future patients.

CTU uses the same scanner machine as CT scans do. The difference between these 2 types of scans is that in addition to collecting the same type of images and information that CT scans do, CTU may also allow the doctor to look at the lining of the tubes that carry urine from the bladder. Looking at the lining of these tubes is something that IVU is used for, and researchers want to find out if CTU can also be used for this purpose.

Study Procedures:

If you are found to be eligible to take part in this study, you will have a CTU procedure performed at least a day before or after your routine IVU. If your doctor has ordered a CT of your abdomen and pelvis and IVU, the CTU will be performed instead of a routine CT scan of the abdomen and pelvis that would normally occur. If your doctor has ordered just a CTU, you will have an IVU as well.

CTU Procedure:

The CTU procedure is very similar to the standard CT of the abdomen/pelvis that you would otherwise receive along with an ITU. To prepare for the CTU, you will be asked to drink contrast solution (a type of dye) in order to allow the tumor(s) to be more easily seen and checked. You will be given about 30 ounces (3 3/4 cups) of contrast solution to drink at 30 minutes before the CTU and another 7 ½ ounces (about a cup) of contrast solution to drink while you are on the scanning table. You will also receive Lasix (furosemide) by injection. Furosemide is given to help the tubes in your kidney dilate (expand) to improve the quality of the images.

For the CTU , you will lie flat on a CT scanner and will receive additional contrast solution by vein during the scan. While the scan is being performed, you will be asked to hold your breath several times, for about 15-20 seconds each time. The process of having the CTU performed should take about 10 minutes longer than a regular CT scan. If the images are not clear enough, all or part of the scanning process may need to be repeated (without repeating the contrast).

IVU Procedure:

Either before the CTU or after it, depending on the order in which you were assigned to receive these procedures, you will receive the IVU as part of your routine care.

Length of Study Participation:

After one set of IVU and CTU scans have been performed, your participation in this study will be over. At least 3 months after your scans are performed, your images will be reviewed a second time by 2 additional M. D. Anderson doctors (radiologists) to compare their findings with the original radiologist's findings.

This is an investigational study. The routine way to check the status of urothelial cancer is to use IVU and CT scanning. It is considered experimental, however, to use CTU instead of routine CT scanning for checking the status of urothelial cancer. At this time, using CTU for this purpose is being done in research only.

Up to 135 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will undergo IVU using digital tomosynthesis and staging abdomino-pelvic CT as part of their routine care will be invited to participate in this study.
2. Patients who have been referred for CTU will also be invited to participate in the study.
3. Such patients will typically

   1. Have histologically proven TCC, or
   2. Have bladder tumors of Stage ≥ T3, or
   3. Had cystectomies for bladder cancer, or
   4. Upper tract TCC.
4. >18 years age.
5. Written informed consent will be obtained from patients.

Patient exclusion criteria:

1. Elevated serum creatinine of >2
2. Allergy to intravenous CT contrast media
3. Ureteral stint present or removed within six weeks
4. Women of child bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2007-11-15 (Actual); Primary Completion 2034-11-30 (Estimated); Study Completion 2034-11-30 (Estimated)

PRIMARY OUTCOMES:
CTU to IVU Technical Performance Comparison: Opacification + Ability to Visualize Urothelial Segments | 2 Years
  Comparison of relative technical performance of computed tomography urography (CTU) to intravenous urography (IVU) using digital tomosynthesis, in terms of visualization and diagnostic quality of segments of the upper urinary tract.

CONTACTS AND LOCATIONS:
Overall Officials: Chaan Ng, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org